CLINICAL TRIAL: NCT00157950
Title: An Immunogenicity and Safety Study of Gardasil (V501 (Human Papillomavirus [Types 6, 11, 16, 18] Recombinant Vaccine)) in Females 9 to 23 Years of Age in Korea
Brief Title: Human Papillomavirus (HPV) Registration Study (Gardasil)(V501-023)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-023; 2005_066
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2010-09-14 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Papillomavirus Infections
Keywords: Human Papilloma Virus
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Gardasil™ (Experimental): Gardasil™ 3 dose regimen
  Interventions: Biological: Gardasil™
- Placebo (Placebo Comparator): Gardasil™ matching placebo 3 dose regimen
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Gardasil™ — Gardasil™ 3 dose regimen (Day 1, Month 2 and Month 6)
  Other Names: V501
  Arms: Gardasil™
Biological: Placebo — Gardasil™ matching placebo 3 dose regimen (Day 1, Month 2 and Month 6)
  Arms: Placebo

SUMMARY:
This is an immunogenicity and safety study of Gardasil (V501) in females 9 to 23 years of age in Korea.

ELIGIBILITY:
Inclusion Criteria:

* Girls ages 9 to 15 years (must not yet have had coitarche)
* Healthy females ages 16 to 23 years (individuals with a lifetime history of 0 to 3 male or female sexual partners)

Exclusion Criteria:

All Subjects:

* History of known prior vaccination with an HPV vaccine.

Women Ages 16 to 23 Only:

* Individuals with any prior history of genital warts or treatment for genital warts.
* Individuals with > 3 lifetime male or female sexual partners.

Ages: 9 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Kang S, Kim KH, Kim YT, Kim YT, Kim JH, Song YS, Shin SH, Ryu HS, Han JW, Kang JH, Park SY. Safety and immunogenicity of a vaccine targeting human papillomavirus types 6, 11, 16 and 18: a randomized, placebo-controlled trial in 176 Korean subjects. Int J Gynecol Cancer. 2008 Sep-Oct;18(5):1013-9. doi: 10.1111/j.1525-1438.2007.01123.x. Epub 2007 Nov 6. PMID 17986242
- [Derived] Hurt L, Nsouli-Maktabi H, Rohrbeck P, Clark LL. Use of quadrivalent human papillomavirus vaccine and the prevalence of antibodies to vaccine-targeted strains among female service members before and after vaccination. MSMR. 2016 Feb;23(2):6-13. PMID 26930146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 10 medical sites in Korea.
  First Patient Treated: 20-Oct-2005
  Last Patient Treated: 24-Jun-2006
Pre-assignment Details: A serum or urine pregnancy test was performed prior to each injection on all subjects. Results were available prior to vaccination. Any subject with a positive pregnancy test at Day 1 was not randomized or vaccinated, and was not eligible to continue in the study.
Period: Overall Study
Arm/Group | Gardasil™ | Placebo
Started | 117 | 59
Vaccinated at Dose 1 | 117 | 59
Vaccinated at Dose 2 | 117 | 59
Vaccinated at Dose 3 | 116 | 59
Completed | 116 | 59
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gardasil™ | Placebo | Total
Number analyzed (Participants) | 117 | 59 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (4.9) | 16.5 (5.2) | 16.6 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 59 | 176
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] | 117 | 59 | 176

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Seroconvert to HPV 6.
Description: Vaccine-induced anti-HPV 6 seroconversion following administration of a 3-dose regimen of GARDASIL® in females 9 to 23 years of age in Korea. Seroconversion for HPV 6 was defined as achieving an anti-HPV cLIA (Competitive Luminex immunoassay) level of at least 20 mMU/mL.
Time Frame: Week 4 Postdose 3
Population: Per-protocol population: subjects must have no major protocol violations, must be seronegative at baseline to the relevant HPV type, and must have post-vaccination data.
Measure: Number; unit: Participants
Arm/Group | Gardasil™ | Placebo
Number analyzed (Participants) | 111 | 58
Participants | 109 | 0
Statistical Analysis 1: Comparison: Gardasil™; Test type: Superiority or Other; Proportion = 98.2, 95% CI 2-sided [93.6 to 99.8] — Exact binomial confidence interval

2. Primary Outcome: Number of Participants Who Seroconvert to HPV 11.
Description: Vaccine-induced anti-HPV 11 seroconversion following administration of a 3-dose regimen of GARDASIL® in females 9 to 23 years of age in Korea. Seroconversion for HPV 11 was defined as achieving an anti-HPV cLIA (Competitive Luminex immunoassay) level of at least 16 mMU/mL.
Time Frame: Week 4 Postdose 3
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gardasil™ | Placebo
Number analyzed (Participants) | 112 | 58
Participants | 112 | 1
Statistical Analysis 1: Comparison: Gardasil™; Test type: Non-Inferiority or Equivalence — The lower bound of the 95% confidence interval for the proportion of subjects receiving Gardasil who were seropositive at Week 4 postdose 3 must be greater than 90%; Proportion = 100, 95% CI 2-sided [96.8 to 100] — Exact binomial confidence interval

3. Primary Outcome: Number of Participants Who Seroconvert to HPV 16.
Description: Vaccine-induced anti-HPV 16 seroconversion following administration of a 3-dose regimen of GARDASIL® in females 9 to 23 years of age in Korea. Seroconversion for HPV 16 was defined as achieving an anti-HPV cLIA (Competitive Luminex immunoassay) level of at least 20 mMU/mL.
Time Frame: Week 4 Postdose 3
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gardasil™ | Placebo
Number analyzed (Participants) | 113 | 58
Participants | 112 | 0
Statistical Analysis 1: Comparison: Gardasil™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Proportion = 99.1, 95% CI 2-sided [95.2 to 100] — Exact binomial confidence interval

4. Primary Outcome: Number of Participants Who Seroconvert to HPV 18.
Description: Vaccine-induced anti-HPV 18 seroconversion following administration of a 3-dose regimen of GARDASIL® in females 9 to 23 years of age in Korea. Seroconversion for HPV 18 was defined as achieving an anti-HPV cLIA (Competitive Luminex immunoassay) level of at least 24 mMU/mL.
Time Frame: Week 4 Postdose 3
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Gardasil™ | Placebo
Number analyzed (Participants) | 110 | 58
Participants | 109 | 0
Statistical Analysis 1: Comparison: Gardasil™; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Proportion = 99.1, 95% CI 2-sided [95.0 to 100] — Exact binomial confidence interval

5. Secondary Outcome: Number of Participants With Adverse Experiences
Description: Number of participants who reported 1 or more adverse experience.
Time Frame: Overall study including 14 calendar days after the last vaccination visit.
Population: All participants who received at least 1 dose of injection.
Measure: Number; unit: Participants
Arm/Group | Gardasil™ | Placebo
Number analyzed (Participants) | 117 | 59
Participants
  Discontinued due to an Adverse Experience (AE) | 0 | 0
  Discontinued due to vaccine related AE | 0 | 0
  Discontinued due to an Serious AE | 0 | 0
  Discontinued due to serious vaccine-related AE | 0 | 0

ADVERSE EVENTS:
Time Frame: During the double-blind period including 14 calendar days after the last vaccination visit.
Description: Although a participant may have had two or more adverse experiences the participant is counted only once in a category. The same participant may appear in different categories.
Arm/Group | Gardasil™ | Placebo
Serious Adverse Events (participants affected / at risk) | 1/117 | 1/59
Other Adverse Events (participants affected / at risk) | 88/117 | 41/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gardasil™ (N=117) | Placebo (N=59)
Traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Acute pharyngitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gardasil™ (N=117) | Placebo (N=59)
Injection site erythema (General disorders) | 27 | 4
Injection site pain (General disorders) | 85 | 30
Injection site swelling (General disorders) | 33 | 7
Injection site tenderness (General disorders) | 2 | 3
Fever (General disorders) | 16 | 10
Cold (Infections and infestations) | 10 | 10
Headache (Nervous system disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.